CLINICAL TRIAL: NCT01293786
Title: Comparison of Vascular Calcification Between Kidney Transplant Recipients and Predialysis Chronic Kidney Disease and Its Association With Serum Magnesium
Brief Title: Serum Magnesium and Vascular Calcification
Status: Completed | Type: Observational
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Sinee Disthabanchong, MD, Division of Nephrology, Department of Medicine, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand
Other Study IDs: 03-02-2011
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2011-05-26 (Estimated); Status verified 2011-05

CONDITIONS: Vascular Calcification; Chronic Kidney Disease
Keywords: magnesium; kidney transplantation; hypomagnesemia
MeSH Terms: conditions — Vascular Calcification; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Kidney transplant recipients
- Chronic kidney disease

SUMMARY:
Both Kidney transplantation (KT) and Chronic Kidney Disease (CKD) patients have reduced kidney function. Low serum magnesium is more prevalent in KT recipients. The present study examines the difference in vascular calcification between KT and CKD and its association with serum magnesium.

DETAILED DESCRIPTION:
Kidney transplantation (KT) improved quality of life and longevity of CKD patients. Nevertheless, kidney function deteriorates overtime in a manner not different from CKD counterparts. Hypomagnesemia is prevalent in KT recipients secondary to immunosuppressive therapy. In addition to serum calcium, phosphate and elemental calcium intake, the relationship between low serum magnesium and vascular calcification (VC) has been observed in small studies in CKD. Whether low serum magnesium associates with VC in KT has never been elucidated. The present study compares vascular calcification between KT and CKD and its association with serum magnesium.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant recipients at least 1 year post surgery
* predialysis chronic kidney disease with serum creatinine > 1.1 mg/dL in female and 1.3 mg/dL in male

Exclusion Criteria:

* acute kidney injury
* parathyroidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients and predialysis chronic kidney disease patients from outpatient nephrology clinic of Ramathibodi hospital, Mahidol University
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The difference in vascular calcification score between KT and CKD | Baseline

SECONDARY OUTCOMES:
The association of serum magnesium with vascular calcification in KT | Baseline
The association of serum magnesium with vascular calcification in CKD | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sinee Disthabanchong, MD, Principal Investigator — Ramathibodi Hospital, Mahidol University
Locations (1):
- Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Phayathai, Bangkok, Thailand